CLINICAL TRIAL: NCT00855647
Title: Hypofractionated Radiotherapy for Localized Prostate Cancer (With CyberKnife or With IMRT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Christopher R. King, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-11022007-792; 79432; NCT00855647; PROS0020
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: Hypo-fractionated Radiotherapy

SUMMARY:
To demonstrate that a hypo-fractionated course of radiotherapy (ie. an accelerated radiotherapy course where fewer but larger doses of radiotherapy are given) is both safe and effective in the treatment of low-risk localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:- Eligible patients will have clinical stage T1c through T2b, initial PSA level <10 and a biopsy Gleason score of 3+3 or 3+4 with fewer than 50% of biopsy cores involved.

* Patients who have had any form of prior curative treatment (surgery, radiotherapy, cryotherapy) will not be eligible. A prior course of hormone therapy of less than 3 months duration will be allowed.
* Adult men will be considered.
* No life expectancy restrictions will apply.
* Performance Status will not be considered.
* No requirements for organ or marrow function will be made
* Ability to understand and the willingness to sign a written informed consent document. Exclusion Criteria:- No prior prostate treatment will be allowed.
* The use of other concurrent Investigational Agents will not be allowed.
* No exclusion requirements due to co-morbid disease or incurrent illness.
* No requirements regarding history of allergic reactions.
* Pregnancy or nursing patients is not applicable (ie. patients are male).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99999 (Estimated)
Dates: Start 2003-08; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
PSA response that achieves a stable nadir over time.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. King, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States